CLINICAL TRIAL: NCT01739738
Title: The Impact of Ureteral Stents on Peristalsis
Status: Withdrawn | Type: Observational
Why Stopped: Study did not start
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Other Study IDs: H12-03027
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Kidney Stones; Tumor; Hydronephrosis
Keywords: peristalsis, kidney stones, hydronephrosis, ureteral stent
MeSH Terms: conditions — Kidney Calculi; Neoplasms; Hydronephrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- no Ureteral Stent - control group: non-stented volunteers to receive ultrasound for peristalsis changes detection
- Ureteral stent: patients who receive stent, and to receive ultrasound for peristalsis changes detection in their stented and non-stented ureter
  Interventions: Device: Ureteral Stent

INTERVENTIONS:
Device: Ureteral Stent — patients who need to receive stent as per standard of care
  Groups: Ureteral stent

SUMMARY:
The purpose of the study is to investigate the impact of ureteral stents on the functioning of ureteral peristalsis (normal contractions in the ureteral organ muscle).

DETAILED DESCRIPTION:
Ureteral stents are commonly used in the field of urology to maintain urinary drainage and are inserted into ureters of patients who suffer from kidney stones, urinary tract infections or cancer. Usually the muscle cells of the ureter contract in a coordinated fashion (peristalsis) in order to provide urinary flow from the kidney into the bladder. By inserting a stent these contractions are disrupted, eventually resulting in a loss of peristalsis. This phenomena is accompanied by swelling of the kidney and pain, which are well-known negative side effects of stents. To avoid stent-related morbidity and improve patients care this issue needs to be investigated further. A first step is to analyse the impact of stents on peristalsis and to possibly bring these results into context with hypothesised molecular mechanisms involved in peristalsis.

ELIGIBILITY:
Inclusion Criteria:

1. stone disease
2. localized tumor disease
3. hydronephrosis of unknown ethiology
4. patients who receive a prophylactic stent before a planned operation.

Exclusion Criteria:

1. Patients being septic and in a life-threatening condition before or after stent-insertion
2. patients with tumors in a progressive state that affect the retroperitoneum (contralateral ureter might be affected and can not serve as a control for the stented side)
3. patients with Morbus Ormond (same reason as above)
4. patients requiring ureteral stents bilaterally (same reason as above)
5. long-term stented patients will be excluded as we are interested in evaluating the onset of changes in peristalsis rate which are expected to be most significant in an acute setting.
6. patients with preexisting abnormalities/pathologies of the urinary tract e.g. reflux disease, megaureter or bladder dysfunctions as these will likely affect our results
7. non English-speaking patients will be excluded as they will not be able to understand the letter of consents.

Exclusion criteria for control group:

1. known preexisting pathology in the urinary tract (see above)
2. volunteers who underwent previous surgical procedures on kidney, ureter or bladder within the past 5 years as this may change the starting position of our study
3. patients currently taking an α-blocker (alfuzosin, terazosin, doxazosin, tamsulosin, prazosin) because these medications are known to affect peristalsis
4. patients currently taking calcium channel blocker (verapamil, diltiazem, nifedipine, nicardipine, bepridil, mibefradil) because these medications are known to affect peristalsis

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who require unilateral insertion of a ureteral stent for the following indications will be included in this clinical trial:
  1. stone disease
  2. localized tumor disease
  3. hydronephrosis of unknown ethiology
  4. patients who receive a prophylactic stent before a planned operation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Effect of stent on ureteral peristalsis in stented ureter | before and after stent insertion (approximately 30 minutes)
  before and after stent insertion (approximately 30 minutes)

SECONDARY OUTCOMES:
Effect of stent on ureteral peristalsis in non-stented ureter | 30 minutes (pre and post stenting)
  Effect of stent on ureteral peristalsis in non-stented ureter pre and post stenting

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia/Vancouver General Hospital, Vancouver, British Columbia, Canada